CLINICAL TRIAL: NCT04691622
Title: Adoptive T Lymphocyte Administration for Chronic Norovirus Treatment in Immunocompromised Hosts
Acronym: ATLANTIC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Michael Keller, MD, Children's National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00014658
Record Dates: First submitted 2020-12-28; First posted 2020-12-31 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Viral Infection; Hematopoietic Stem Cell Transplantation (HSCT); Primary Immunodeficiency Disorders (PID)
MeSH Terms: conditions — Virus Diseases; Primary Immunodeficiency Diseases | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Norovirus -specific T-cell (NST) therapy for chronic norovirus infection (Experimental): This is a Phase I dose-escalation study to evaluate the safety of norovirus -specific T-cell (NST) therapy for chronic norovirus infection in participants following hematopoietic stem cell transplantation (HSCT) or with primary immunodeficiency disorders (PID) who have not undergone HSCT. There are two arms in this study:
  1. Arm A: Participants who receive donor-derived NST therapy after HSCT
  2. Arm B: Participants who receive partially HLA matched NSTs. The following participants apply:
     * Participants with PID who have not undergone HSCT.
     * Participants who have undergone HSCT but do not have available donor derived NSTs, or those for whom NSTs cannot be generated due to norovirus seronegativity.
     * Participants who have undergone SOT.
  Interventions: Biological: Norovirus -specific T-cell (NST) therapy

INTERVENTIONS:
Biological: Norovirus -specific T-cell (NST) therapy — Arm A: Investigators will test three doses: 1 x 107 /m2, 2 x 107 /m2, and 4 x 107 /m2. After infusion, participants will have a 45-day safety monitoring period for immediate toxicities following infusion.
  Arm B: Investigators will test three doses: 1 x 107 /m2, 2 x 107 /m2, and 4 x 107 /m2. After infusion, participants will have a 45-day safety monitoring period for immediate toxicities following infusion.

SUMMARY:
This is a Phase I dose-escalation study to evaluate the safety of norovirus -specific T-cell (NST) therapy for chronic norovirus infection in participants following hematopoietic stem cell transplantation (HSCT) or who are immunocompromised due to PID and have not undergone HSCT, or Solid Organ Transplant (SOT) recipients.

DETAILED DESCRIPTION:
This is an open label, phase I study of norovirus-specific T-cell immunotherapy for treatment of participants with primary immunodeficiency disorders (PID) and chronic norovirus. This study is designed to assess the safety of norovirus-specific T-cell (NST) infusion in this population. There are two arms in this study:

1. Arm A: Participants who receive donor derived NST therapy after HSCT
2. Arm B: Participants who receive partially HLA matched NSTs. The following participants apply:

   * Participants with PID who have not undergone HSCT.
   * Participants who have undergone HSCT but do not have available donor derived NSTs, or those for whom NSTs cannot be generated due to norovirus seronegativity.
   * Participants who have undergone SOT.

Participants will be monitored for infusion-related reactions and GVHD for 1 year following first infusion. During this time, participants will be accessed with regard to the length and quantity of norovirus shedding in stool, and gastrointestinal and constitutional symptoms will be scored by clinicians and participants. Correlative studies of T-cell immune reconstitution against norovirus, norovirus genomic sequences, and composition of the fecal microbiome will also be accessed.

The primary purpose of this phase I study is to assess the safety of administering donor-derived or partially HLA-matched NSTs in immunocompromised participants with chronic norovirus infections. Related and unrelated donors of participants who have chronic norovirus infection after HSCT will be enrolled for screening and production of NSTs from peripheral blood. Following product manufacturing, participants who have undergone HSCT (Arm A) will receive donor-derived NSTs. For participants with PID who have not undergone HSCT or recipients of SOT (Arm B), high-resolution HLA typing of the participant will be utilized for an inquiry of the NST bank to determine if a partially HLA-matched NST product exists that has antiviral activity mediated through one or more shared HLA alleles. Participants who have undergone HSCT but either do not have available donors for NST generation, or who have donors from whom NSTs cannot be generated due to norovirus seronegativity will also be eligible for inquiry for treatment with partially HLA-matched NSTs if available under study Arm B.

This will be a dose escalation study with two arms. Participants who have undergone HSCT will be enrolled on Arm A and receive NSTs derived from their HSCT donor. Participants with a diagnosis of PID who have not undergone HSCT, recipients of SOT, or participants who have undergone HSCT but do not have available donor-derived NSTs will be enrolled on Arm B and receive partially HLA-matched NSTs. We will test three doses: 1x107 /m2, 2x107 /m2, and 4x107 /m2. Investigators will have a 45-day safety monitoring period for immediate toxicities following infusion.

ELIGIBILITY:
Inclusion Criteria:

Participant Inclusion Criteria for NST Infusion:

1. Participants must meet one of the following criteria:

   1. Recipient of prior myeloablative or non-myeloablative allogeneic hematopoietic stem cell transplant using either bone marrow or peripheral blood stem cells or single or double cord blood OR
   2. Primary immunodeficiency disorder (as defined by clinical and laboratory evaluations)81 and have not undergone HSCT, OR
   3. Recipients of solid organ transplant.
2. Documentation of chronic norovirus infection:

   a. Chronic norovirus infections will be defined as having consecutive positive norovirus stool tests (2 or more) spanning a minimum three-month period with attributable signs and symptoms of norovirus disease.
3. Participants receiving steroids for treatment of GVHD or for other reasons, dosage must have been tapered to <0.5 mg/kg/day of prednisone (or equivalent) a minimum of 7 days prior to infusion.

   a. Treatment with enteral topical steroids such as Budesonide at standard doses may be continued if previously utilized but should not be newly initiated in the 3 months after NST therapy.
4. For participants who have undergone HSCT, participants must have stable donor chimerism within the 30 days prior to NST infusion.

   a. Stability will be defined as i. >95% donor chimerism in CD33 and/or whole blood chimerism. OR ii. >90% donor chimerism with <5% change between subsequent tests separated by at least 1 week.
5. For recipients of solid organ transplants, participants must have stable graft function on maintenance immunosuppression, without evidence of rejection in the past 2 months prior to infusion, as defined by:

   a. Stability of relevant functional testing in the previous 2 months, defined as: i. Renal transplant: renal function ≥ grade 3 per the National Kidney Foundation K/DOQI Clinical Practice Guidelines for Chronic Kidney Disease (2002) ii. Cardiac transplant: maintenance of LVEF >40% iii. Lung transplant: lack of baseline oxygen requirement iv. Liver transplant: AST/ALT ≤3x upper limit normal and bilirubin ≤2x upper limit normal b. Donor-derived cell free DNA <2x upper limits for assay in the previous 2 months, c. Stable donor-specific antibody profile in the previous 2 months. i. No increase in antibody titers between most recent testing in the previous 2 months and prior testing.
6. Karnofsky/Lansky score >50
7. 3 months to 80 years of age at enrollment.
8. ANC ≥500/ul.
9. Hemoglobin ≥7.0g/dl (level can be achieved with transfusion).
10. Platelets ≥20 K/ul (level can be achieved with transfusion).
11. Bilirubin ≤2x upper limit normal.
12. AST ≤3x upper limit normal.
13. Serum creatinine ≤2x upper limit normal OR estimated GFR ≥30 ml/hr.
14. Pulse oximetry of ≥90% on room air.
15. Negative pregnancy test in female participant of childbearing age.
16. Written informed consent and/or signed assent line from participant, parent or guardian.

Donor Inclusion Criteria:

1. Donors who have fulfilled eligibility as per United States Food and Drug Administration (FDA) regulations outlined in 21 Code of Federal Regulations (CFR) 1271 subpart C. This includes that donors have been deemed in good health by donor physician based on physical examination and laboratory testing. If a donor has been chosen for the transplant based on urgent medical need, that same donor will also be used for NST generation provided that there are no new reasons for ineligibility since the stem cell collection.
2. For third-party banking, donors must be between 2 to 35 years of age (females) or 2 to 40 years of age (males).
3. Donor or guardian of pediatric donor capable of providing informed consent.
4. Donor (related or unrelated) must have completed Infectious Disease (ID) testing up to 7 days before or after the collection of blood for NST manufacturing. The following tests will be performed:

   * HBsAg
   * HBc Antibody
   * HCV Antibody
   * HIV 1/2 Antibody
   * HTLV I/II Antibody
   * T. Cruzi Antibody (Chagas)
   * CMV Total Antibody
   * Syphilis (T. Pallidum IgG and IgM)
   * HBV, HCV, HIV Nucleic Acid testing (NAT)
   * WNV NAT
5. Female donors of childbearing age must have a negative pregnancy test and not be lactating.

Exclusion Criteria:

Participants Exclusion Criteria for NST Infusion:

1. Participants receiving biological or immunosuppressive monoclonal antibodies targeting T cells within 28 days prior to NST infusion, including ATG, Alemtuzumab, Basiliximab, Tocilizumab, Brentuximab, or other medications under this category as determined by the investigators.

   a) If alemtuzumab has been received within 6 weeks prior to NST infusion, plasma levels should be obtained to ensure drug clearance (≤0.16 pg/ml).
2. Participants who have received donor lymphocyte infusion (DLI), chimeric antigen receptor T cell infusion, or other experimental cellular therapies within 28 days prior to NST infusion.
3. Participants with SCID who have undergone α/β TCR depleted HSCT within the past 100 days post-transplant.
4. Participants who have received ruxolitinib or other JAK inhibitors within 7 days prior to NST infusion.
5. Participants with uncontrolled or progressing infections other than norovirus. Uncontrolled infections are defined as bacterial, fungal, or non-targeted viral infections with either clinical signs of worsening despite standard therapy, or chronic gastrointestinal symptoms that may be attributed to the uncontrolled infection. Progressing infection is defined as hemodynamic instability, worsening physical signs, or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.

   1. For bacterial infections, participants must be receiving definitive therapy and have no signs of progressing infection within 7 days prior to NST infusion and or no chronic gastrointestinal symptoms associated with this bacterial infection.
   2. For fungal infections, participants must be receiving definitive systemic anti-fungal therapy and have no signs of progressing infection within 7 days prior to NST infusion.
6. Participants must not have other active gastrointestinal infections to which symptoms may be attributable, including parasitic infections (cryptosporidium, giardiasis), viral infections aside from norovirus (CMV colitis, rotavirus, adenovirus), or bacterial infections with C. difficile, Yersinia, Campylobacter, Salmonella, Shigella, or enteroinvasive or enterotoxigenic E. coli.

   a) Testing for unrelated gastrointestinal (GI) infections must be performed within 14 days prior to NST infusion, and must include: i. Crytosporidium/Giardia testing via antigen or PCR testing. ii. Stool viral testing for rotavirus and adenovirus via antigen or PCR testing.

   iii. Stool bacterial culture or PCR testing. iv. C. difficile toxin PCR. b) Determination of active infection versus chronic carriage/shedding will be made by the investigators and clinical providers and will depend on the presence of clinical symptoms corresponding with the timing of positive test results, presence of a clinical response to targeted therapy, and by histological or other testing if clinically indicated.
7. Participants with active and uncontrolled relapse of malignancy (if applicable).

   1. Failure of primary engraftment is defined as failure to achieve platelet and/or neutrophil engraftment (ANC <500/ul and/or platelets <20 K/ul) following HSCT.
   2. Secondary graft failure is defined as <5% donor chimerism (CD3+ or CD34+) or permanent loss of neutrophil and/or platelet engraftment (ANC <500/ul and/or platelets <20 K/ul) at any time after primary engraftment.
8. Participants with symptomatic gastrointestinal conditions aside from norovirus, including active inflammatory bowel disease or graft versus host disease (grades 2 to 4).
9. Participants who have received a small bowel transplant.
10. Participants receiving checkpoint inhibitors within the previous 3 months prior to NST infusion, including nivolumab, pembrolizumab, or other related medications.
11. For SOT recipients, alteration in immunosuppression as follows:

    1. Any intensification of immunosuppression (including but not limited to pulse dose corticosteroids or new biologic therapies) in the previous 2 months,
    2. Alteration of maintenance immunosuppression (including changes in the number of agents or dosing goals) in the previous month.
12. Participants who have received enteral immunoglobulin, nitazoxanide, or other experimental therapies for norovirus infection within 28 days prior to NST infusion.
13. Co-enrollment in other trials is restricted, other than enrollment on natural history or observational studies. Study staff should be notified of co-enrollment as it may require the approval of the investigator or sponsor.

Donor Exclusion Criteria:

1. Donation of cells would pose a physical or psychological risk to the donor

Ages: 3 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-03-17 (Actual); Primary Completion 2028-08-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute GvHD (grade III-IV) | Within 45 days of first NSTs infusion
  Number of patients with acute GvHD grades III-IV
Incidence of infusion related adverse events as per CTCAE common criteria guidelines. | Within 45 days of first NSTs infusion
  Number of patients with Grades 3-5 infusion-related adverse events
Incidence of non-hematological adverse events | Within 45 days of first NSTs infusion
  Number of patients with Grades 4-5 non-hematological adverse events related to the NST product within 45 days of the first infusion

SECONDARY OUTCOMES:
Antiviral activity | Stool viral loads will be evaluated for 12 months following the final NST infusion.
  Antiviral activity will determined by measurements in viral loads by RT-PCR from stool samples in comparison to the mean baseline viral load.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Keller, MD, Principal Investigator — CNH
Locations (3):
- United States (3):
  - Children's National Hospital, Washington D.C., District of Columbia
  - Johns Hopkins University, Baltimore, Maryland
  - National Institutes of Health (NIH), Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No
Data will be made available via publication. All raw data, methodologies and statistical analyses will also be made available upon publication.